CLINICAL TRIAL: NCT02332278
Title: Early Oral Feeding Versus Traditional Postoperative Care After Uncomplicated Cesarean Section. A Randomized Controlled Trial.
Brief Title: Early Oral Feeding Versus Traditional Postoperative Care After Cesarean Section.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Thomas Hospital, Panama (Other)
Responsible Party: Principal Investigator, Osvaldo A. Reyes T., Coordinator of research, Saint Thomas Hospital, Panama
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MHST2014-08
Record Dates: First submitted 2015-01-04; First posted 2015-01-06 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2015-01

CONDITIONS: Complications; Cesarean Section
Keywords: Cesarean section; Early feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early feeding (Experimental): Early feeding (fluid diet), four hours after cesarean section.
  Interventions: Procedure: Early feeding
- Late feeding (Active Comparator): Late feeding (fluid diet) 12 hours after cesarean section.
  Interventions: Procedure: Late feeding

INTERVENTIONS:
Procedure: Early feeding — Fluid diet four hours after cesarean section
  Arms: Early feeding
Procedure: Late feeding — Fluid diet 12 hours after cesarean section
  Arms: Late feeding

SUMMARY:
To determine the effect in the post operative period of early feeding (4 hours after surgery) vs. traditional management (feeding 12 hours after surgery) in uncomplicated cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Cesarean section with regional anesthesia, regardless of gestational age.

Exclusion Criteria:

* Use of magnesium sulphate
* General anesthesia
* Pre gestational or gestational diabetes
* Bowel injury during surgery

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 444 (Actual)
Dates: Start 2014-06; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Adynamic ileus | 72 hours
  Presence of signs of adynamic ileus (nausea, vomiting, abdominal distention) after feeding

SECONDARY OUTCOMES:
Post operative pain | 72 hours
  Level of pain, using a visual scale (12, 24, 48 and 72 hours after surgery)
Satisfaction | 72 hours
  Personal satisfaction, using a numeric scale (12, 24, 48 and 72 hours after surgery)

CONTACTS AND LOCATIONS:
Overall Officials: Ana Lia Becerra, MD, Principal Investigator — Saint Thomas Hospital, Panama; Osvaldo Reyes, MD, Principal Investigator — Saint Thomas Hospital, Panama
Locations (1):
- Saint Thomas H, Panama City, Provincia de Panamá, Panama